CLINICAL TRIAL: NCT04079205
Title: Home-based Rehabilitation Using Smart Wearable Knee Exercise Device With Electrical Stimulation After Anterior Cruciate Ligament Reconstruction: A Study Protocol for a Randomized Controlled Trial
Brief Title: Home Rehabilitation Using Smart Wearable Exercise and Electrical Stimulation Device After Anterior Cruciate Ligament Reconstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulty in patient enrollment
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Ministry of SMEs and Startups, Korea (Unknown); Exosystems CO.,Ltd (Unknown)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-1806-475-006
Record Dates: First submitted 2019-05-08; First posted 2019-09-06 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Anterior Cruciate Ligament Reconstruction; Wearable device; Knee; Neuromuscular Electrical Stimulation; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home rehabilitation using Wearable Device (Experimental): Home rehabilitation using Wearable Device(exoRehab)
  Interventions: Device: Wearable Device(exoRehab)
- Control (Active Comparator): Standard home rehabilitation program
  Interventions: Behavioral: Home rehabilitation program

INTERVENTIONS:
Device: Wearable Device(exoRehab) — rehabilitation program for patients after Anterior Cruciate Ligament Reconstruction using Wearable Device (exoRehab)
  Arms: Home rehabilitation using Wearable Device
Behavioral: Home rehabilitation program — rehabilitation program for patients after Anterior Cruciate Ligament Reconstruction
  Arms: Control

SUMMARY:
The purpose of this study is to develop and apply a rehabilitation program for patients who are discharged after ACL reconstruction using a wearable joint rehabilitation exercise device (exoRehab).

DETAILED DESCRIPTION:
This randomized, single-blind, controlled trial included 40 patients who are discharged after ACL reconstruction.

The intervention group(n=20) was instructed and educated about 6 week home rehabilitation program using a wearable device(exoRehab)

The controls(n=20) was instructed and educated about 6 week conventional home rehabilitation program

Two weeks after surgery and six weeks after discharge, evaluation is performed.

The purpose of this study is to develop and apply a rehabilitation program for patients who are discharged after ACL reconstruction using a wearable joint rehabilitation exercise device (exoRehab).

ELIGIBILITY:
Inclusion Criteria:

* Patients with anterior cruciate ligament reconstruction
* Patients who are older than 19 years of age

Exclusion Criteria:

* History of surgery or traumatic injury to the uninvolved lower extremity
* Complication after ACL reconstruction surgery
* Dermatological conditions affecting the thigh
* Body mass index (BMI) greater than 40 kg/m2
* Implanted pacemakers or defibrillators
* Significant neurologic impairments
* Other unstable lower-extremity orthopedic conditions
* Initiated rehabilitation at another facility prior to their first physical therapy session at our facility
* Other lower limb impairment affecting function
* More than one surgery for a tear of the ACL

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle strength using dynamometry | Baseline and 6 weeks
  Change from baseline quadriceps muscle strength at 6 weeks

SECONDARY OUTCOMES:
Active range of motion of knee | Baseline, 2 weeks and 6 weeks
  Change from baseline active range of motion of knee at 2 weeks and 6 weeks
Passive range of motion of knee | Baseline, 2 weeks and 6 weeks
  Change from baseline passive range of motion of knee at 2 and 6 weeks
Root mean square of surface electromyography of quadriceps muscle | Baseline, 2 weeks and 6 weeks
  Change from baseline root mean square of surface electromyography of quadriceps muscle at 2 weeks and 6 weeks
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Score | Baseline, 2 weeks and 6 weeks
  Changes from baseline in International Knee Documentation Committee (IKDC) subjective score at 2 weeks and 6 weeks, Higher scores indicate better recovery
Lysholm score | Baseline, 2 weeks and 6 weeks
  Change from baseline in Lysholm score at 2 weeks and 6 weeks. Lysholm score ranges from 0-100 with higher scores indicating better knee joint function.
Knee Outcome Survey-Activities of Daily Living Scale | Baseline, 2 weeks and 6 weeks
  Change from baseline in score of Knee Outcome Survey-Activities of Daily Living Scale at 2 weeks and 6 weeks. Score ranges from 0-100 with higher scores indicating better knee joint function.
EQ-5D-3L Scores | Baseline, 2 weeks and 6 weeks
  Change from baseline in EQ-5D-3L Scores at 2 weeks and 6 weeks. EQ-5D-3L is made up for two components. First, the health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; each dimension ranging from 1-3. From these five dimensions, EQ-5D index is calculated, having a value between 0-1. Second, the evaluation part involves an analogue scale, asking to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. Zero corresponds to " the worst health you can imagine", and hundred corresponds to "the best health you can imagine".
Visual Analogue Scale for pain | Baseline, 2 weeks and 6 weeks
  Change from baseline in Visual Analogue Scale at 2 weeks and 6 weeks. The Visual Analogue Scale(VAS), a 101-point scale for evaluating pain which consists of a 100-millimetre scale ranging from 0 (no pain at all) to 100 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, Ph.D, Principal Investigator — Seoul National University Bundang Hospital, Seongnam, South Korea
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim G, Kim WS, Kim TW, Lee YS, Lee H, Paik NJ. Home-based rehabilitation using smart wearable knee exercise device with electrical stimulation after anterior cruciate ligament reconstruction: A study protocol for a randomized controlled trial. Medicine (Baltimore). 2020 May;99(20):e20256. doi: 10.1097/MD.0000000000020256. PMID 32443364